CLINICAL TRIAL: NCT06091969
Title: Nutraceutical Supplementation for Male Subfertility
Brief Title: Supplementation for Male Subfertility
Acronym: FertEnhancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: One Fertility (Other)
Responsible Party: Principal Investigator, Mark Tarnopolsky, Professor, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16502
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Male Infertility
Keywords: Sub-fertility; Infertility; Antioxidants; Supplements; Creatine; Arginine; Vitamins; Aging; Oxidative stress; Inflammation; DNA; Mitochondria; Fragmentation; ATP; Weight loss; Obesity
MeSH Terms: conditions — Infertility, Male; Infertility; Inflammation; Weight Loss; Obesity

STUDY DESIGN:
Intervention Model Description: This is a 3-month placebo-controlled, double-blinded, randomized clinical trial comparing an active supplement designed to enhance sperm function (Fertility Enhancer) to an inactive placebo (PLACEBO) in overweight or obese and subfertile males.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Volunteers will be given an identifier number and then randomized into placebo or active groups by an independent third party meaning that all participants, care providers and investigators will be blinded to the treatment allocations until the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active multi-ingredient supplement (Fertility Enhancer; FE) (Experimental): Volunteers will be randomized in a double-blinded fashion into the experimental treatment group, which entails daily supplementation of an active multi-ingredient supplement designed to enhance fertility (Fertility Enhancer; FE) for 3 months.
  Interventions: Dietary Supplement: Active multi-ingredient supplement (Fertility Enhancer, FE)
- Inactive placebo (Placebo; PLA) (Placebo Comparator): Volunteers will be randomized in a double-blinded fashion into a placebo group, which entails daily supplementation of a calorie-matched, inactive placebo (Placebo; PLA) identical in flavor to the active supplement for 3 months.
  Interventions: Dietary Supplement: Inactive placebo (Placebo; PLA)

INTERVENTIONS:
Dietary Supplement: Active multi-ingredient supplement (Fertility Enhancer, FE) — Consuming a multi-ingredient supplement targeting multiple cell pathways daily for 3 months.
  Arms: Active multi-ingredient supplement (Fertility Enhancer; FE)
Dietary Supplement: Inactive placebo (Placebo; PLA) — Consuming an inactive placebo that is calorie-matched to the active supplement daily for 3 months.
  Arms: Inactive placebo (Placebo; PLA)

SUMMARY:
Old age, obesity, physical inactivity, environmental factors and genetics may contribute negatively to fertility in both males and females. In males, specifically, certain supplements, such as single antioxidants and trace minerals, have previously been shown to improve sperm function marginally. One hypothesis is that sperm function can be improved even further by combining several different types of supplements (e.g., amino acids, energy carriers, vitamins, antioxidants, and trace minerals) to target several age-related cell pathways, for example, oxidative stress, mitochondrial dysfunction, inflammation and cell energetics. This 3-month placebo-controlled, randomized clinical trial, aims to test the effects of a novel multi-ingredient supplement (Fertility Enhancer) that targets several age-related cell pathways on sperm function in overweight or obese and subfertile males.

DETAILED DESCRIPTION:
BACKGROUND: Infertility is characterized by the failure to become pregnant after one year of regular intercourse without the use of contraceptives and impacts 10-15% of couples worldwide. Both male and female partners contribute to a couple's reproductive health, with approximately one third of infertility cases caused by male factors, one third by female factors, and the remaining by either a combination of both or unknown causes. The prevalence of infertility is a growing concern in Canada, as is seen in an increased use of assisted reproductive technology (ART), which may be both invasive and expensive. Cost-effective, safe, and accessible alternatives to ART are therefore needed. The most common cause of subfertility is 'biological aging', characterized by the hallmarks of aging, such as mitochondrial dysfunction, oxidative damage and inflammation. Another common cause of male and female subfertility is obesity, which is associated with multisystemic oxidative damage and inflammation.

PURPOSE: The aim of this placebo-controlled, double-blind randomized clinical trial is to test the effects of a multi-ingredient supplement (Fertility Enhancer) designed to target several aging- and obesity-related pathways on World Health Organization (WHO) semen quality parameters in overweight and obese and subfertile males (sperm count, motility, morphology and vitality).

SAMPLE-SIZE ESTIMATE AND DESIGN: Sperm count/concentration is strongly correlated to all World Health Organization semen quality parameters. With significance set at 0.05 (Z = 1.96) and power to 0.8 (Z = 0.84), a sample-size of 17-32 per group is sufficient to detect an increase of 10 x 10^6 spermatozoa/mL with a standard deviation of 15 to 20 x 10^6 spermatozoa/mL. Thus, sixty-four (n = 64) males between 25 and 50 years of age that are confirmed overweight or obese and subfertile will be randomized into age-matched Placebo (PLA, n = 32) vs Fertility Enhancer (FE, n = 32) groups and undergo daily supplementation for 3 months.

SUPPLEMENTS: The FE supplement contains energy carriers (creatine), conditionally essential amino acids (arginine), Omega 3 fatty acids (DHA and EPA), vitamins (B9, B12, E, and D3), antioxidants (CoQ10 and alpha lipoic acid), trace minerals (selenium, iron, zinc, and copper), and plant extracts (beet root, green tea, and green coffee bean). The isocaloric and inactive placebo contains safflower oil, microcrystalline cellulose and sugar and is identical in flavor to FE.

CO-PRIMARY OUTCOMES: All outcomes will be measured at baseline and post intervention for assessing % pre-to-post changes. Co-primary outcomes are body composition by dual x-ray absorptiometry, including lean mass to fat mass ratio (body composition index; BCI) and total fat mass, and the WHO semen quality parameters; specifically, % improvements in sperm count, motility, morphology, and vitality.

SECONDARY OUTCOMES: Secondary outcomes are % improvements in sperm DNA fragmentation (flow cytometry-assessed) and markers of oxidative damage (protein carbonyls, lipid peroxidation, 8-hydroxydeoxyguanosine)), inflammation (interleukin-1, tumor necrosis factor-alpha, interleukin-6), apoptosis (total and cleaved caspase 3), cell cycle arrest (p16 and p21), mitochondrial biogenesis (complexes I-V), antioxidant status (superoxide dismutases 1 and 2), and energy state (ATP and phosphocreatine).

OTHER: Additional outcomes are body morphology (bodyweight, waist/height ratio, and body mass index), other body composition outcomes (lean mass and appendicular skeletal muscle mass index), and blood markers of oxidative damage (malondialdehyde), inflammation (c-reactive protein, interleukin-1, tumor necrosis factor-alpha, interleukin-6), antioxidant status (ORAC, TEAC), liver enzymes (alanine aminotransferase, aspartate aminotransferase, and creatinine) and energy state (ATP & phosphocreatine levels).

HYPOTHESIS: The main hypothesis of the current trial is that co-primary body composition outcomes and the World Health Organization (WHO) semen quality parameters (count, motility, morphology, and/or vitality) will be significantly improved following FE supplementation and superior to PLA.

STATISTICS: A standard omnibus one-way repeated measures ANOVA F-test followed by Duncan post hoc analyses will be used for all parametric data analyses. Non-parametric equivalents will be used for non-normally distributed data with significance set at p = 0.05. Delta pre-post changes (% improvements) for all outcomes within and between groups are biologically relevant and planned a priori comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Males between the ages of 25-50 years diagnosed with subfertility through Ontario Networks of Experts in Fertility (ONE Fertility, Burlington, ON).
* For diagnosis of male subfertility, the 2010 and 2021 World Health Organization criteria will be used for sperm count, motility, morphology and vitality.
* Overweight and obese males according to body mass index (BMI) between the ages of 25-50 years.

Exclusion Criteria:

* Smoking,
* history and drug alcohol abuse,
* BMI > 30 kg/m2,
* genital disease (cryptorchidism, current genital inflammation, or varicocele),
* genital trauma or surgery to the male reproductive system,
* known Y chromosome microdeletions or karyotype abnormalities (if known prior),
* hepatobiliary disease,
* significant renal insufficiency,
* occupational exposures to reproductive toxins,
* endocrine abnormality,
* recent or current sexually transmitted infection,
* use of cytotoxic drugs,
* use of immunosuppressants,
* use of anticonvulsants,
* use of androgens or antiandrogens,
* history of central nervous system injury,
* neurological or psychiatric disease to potentially compromise study data collection,
* treatment of erectile dysfunction with any drugs during the past 4 weeks,
* history of cancer chemotherapy,
* current supplementation with ingredients being tested unless 1-month washout period

Ages: 25 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-02-02 (Estimated); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
Percent change in body composition index from baseline to 3 months | Baseline to 3 months
  Lean mass/fat mass ratio by dual X-ray absorptiometry scan (body composition index; % change)
Percent change in total fat mass from baseline to 3 months | Baseline to 3 months
  Total fat mass by dual X-ray absorptiometry scan (kg; % change)
Percent change in sperm count/concentration from baseline to 3 months | Baseline to 3 months
  Sperm count/concentration (millions spermatozoa/mL semen)
Percent change in sperm motility from baseline to 3 months | Baseline to 3 months
  Proportion motile sperm (%)
Percent change in sperm morphology from baseline to 3 months | Baseline to 3 months
  Proportion normal sperm morphology (%)
Percent change in sperm vitality from baseline to 3 months | Baseline to 3 months
  Proportion viable sperm (vitality) (%)

SECONDARY OUTCOMES:
Percent change in sperm DNA fragmentation index from baseline to 3 months | Baseline to 3 months
  Sperm DNA fragmentation index by flow cytometry (%)
Percent change in sperm DNA 8-hydroxydeoxyguanosine from baseline to 3 months | Baseline to 3 months
  Sperm DNA 8-hydroxydeoxyguanosine by ELISA (ng/mL; %)
Percent change in sperm protein carbonyls from baseline to 3 months | Baseline to 3 months
  Sperm protein carbonyls immunoblot (optical density; %)
Percent change in sperm lipid peroxidation (4-hydroxynonenal) from baseline to 3 months | Baseline to 3 months
  Sperm 4-hydroxynonenal immunoblot (optical density; %)
Percent change in sperm antioxidant marker superoxide dismutase 1 from baseline to 3 months | Baseline to 3 months
  Sperm superoxide dismutase 1 expression immunoblot (optical density; %)
Percent change in sperm antioxidant marker superoxide dismutase 2 from baseline to 3 months | Baseline to 3 months
  Sperm superoxide dismutase 2 expression immunoblot (optical density; %)
Percent change in sperm apoptotic marker cleaved caspase 3 from baseline to 3 months | Baseline to 3 months
  Sperm cleaved caspase 3 expression immunoblot (optical density; %)
Percent change in sperm apoptotic marker total caspase 3 from baseline to 3 months | Baseline to 3 months
  Sperm total caspase 3 expression immunoblot (optical density; %)
Percent change in sperm mitochondrial OXPHOS from baseline to 3 months | Baseline to 3 months
  Sperm mitochondrial OXPHOS expression immunoblot (optical density; %)
Percent change in sperm cell cycle arrest marker p16 from baseline to 3 months | Baseline to 3 months
  Sperm p16 messenger RNA levels by rtPCR (fold control/placebo; %)
Percent change in sperm cell cycle arrest marker p21 from baseline to 3 months | Baseline to 3 months
  Sperm p21 messenger RNA levels by rtPCR (fold control/placebo; %)
Percent change in sperm inflammatory marker interleukin 1 from baseline to 3 months | Baseline to 3 months
  Sperm interleukin 1 messenger RNA levels by rtPCR (fold control/placebo; %)
Percent change in sperm inflammatory marker TNF-alpha from baseline to 3 months | Baseline to 3 months
  Sperm TNF-alpha messenger RNA levels by rtPCR (fold control/placebo; %)
Percent change in sperm inflammatory marker interleukin-6 from baseline to 3 months | Baseline to 3 months
  Sperm interleukin-6 messenger RNA levels by rtPCR (fold control/placebo; %)
Percent change in sperm inflammatory marker interleukin-8 from baseline to 3 months | Baseline to 3 months
  Sperm interleukin-8 messenger RNA levels by rtPCR (fold control/placebo; %)
Percent change in sperm inflammatory marker interleukin-18 from baseline to 3 months | Baseline to 3 months
  Sperm interleukin-18 messenger RNA levels by rtPCR (fold control/placebo; %)
Percent change in sperm inflammasome marker caspase 1 from baseline to 3 months | Baseline to 3 months
  Sperm caspase 1 messenger RNA levels by rtPCR (fold control/placebo; %)
Percent change in sperm ATP levels from baseline to 3 months | Baseline to 3 months
  Sperm ATP levels by ELISA (pM/100 mg protein; %)
Percent change in sperm phosphocreatine levels from baseline to 3 months | Baseline to 3 months
  Sperm phosphocreatine levels by ELISA (ng/100 mg protein; %)

OTHER OUTCOMES:
Percent change in bodyweight from baseline to 3 months | Baseline to 3 months
  Bodyweight by standard scale (kg; %)
Percent change in body mass index from baseline to 3 months | Baseline to 3 months
  Body mass index (BMI) (bodyweight/height squared; kg/m2; %)
Percent change in lean mass from baseline to 3 months | Baseline to 3 months
  Lean mass by dual X-ray absorptiometry scan (kg; %)
Percent change in appendicular skeletal muscle mass from baseline to 3 months | Baseline to 3 months
  Appendicular skeletal muscle mass by dual X-ray absorptiometry scan (kg; %)
Percent change in appendicular skeletal muscle mass index from baseline to 3 months | Baseline to 3 months
  Appendicular skeletal muscle mass index by dual X-ray absorptiometry scan (kg/height squared; %)
Percent change in liver enzyme ALT from baseline to 3 months | Baseline to 3 months
  Serum alanine aminotransferase levels (IU/L; %)
Percent change in liver enzyme AST from baseline to 3 months | Baseline to 3 months
  Serum aspartate aminotransferase levels (IU/L; %)
Percent change in liver enzyme creatinine from baseline to 3 months | Baseline to 3 months
  Serum creatinine levels (mg/dL; %)
Percent change in malondialdehyde levels from baseline to 3 months | Baseline to 3 months
  Plasma malondialdehyde levels (uM; %)
Percent change in Oxygen Radical Absorbance Levels (ORAC) from baseline to 3 months | Baseline to 3 months
  Plasma Oxygen Radical Absorbance Levels (ORAC units; %)
Percent change in Trolox Equivalent Antioxidant Capacity (TEAC) from baseline to 3 months | Baseline to 3 months
  Serum Trolox Equivalent Antioxidant Capacity (mM; %)
Percent change in inflammatory cytokine interleukin-1 from baseline to 3 months | Baseline to 3 months
  Serum interleukin 1 levels (pg/mL; %)
Percent change in inflammatory cytokine interleukin-6 from baseline to 3 months | Baseline to 3 months
  Serum interleukin-6 levels (pg/mL; %)
Percent change in inflammatory cytokine TNF-alpha from baseline to 3 months | Baseline to 3 months
  Serum TNF-alpha levels (pg/mL)
Percent change in inflammatory marker c-reactive protein from baseline to 3 months | Baseline to 3 months
  Serum c-reactive protein levels (mg/dL; %)
Percent change in ATP levels from baseline to 3 months | Baseline to 3 months
  Plasma ATP levels (mmol/L; %)
Percent change in phosphocreatine levels from baseline to 3 months | Baseline to 3 months
  Plasma phosphocreatine levels (mmol/L; %)

CONTACTS AND LOCATIONS:
Locations (1):
- Mark Tarnopololsky, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, informed consent form and statistical analysis plan may be made available from February 2025 onward. This may occur along with the release of the deidentified results for publishing requirements and/or upon request by qualified researchers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study protocol, informed consent form and statistical analysis plan may be made available from February 2025 onward. This may occur along with the release of the deidentified results for publishing requirements and/or upon request by qualified researchers.
Access Criteria: Access to trial data can be requested by qualified researchers engaging in independent scientific research studies.